CLINICAL TRIAL: NCT00305708
Title: Bone Marrow Stem Cell Transplantation for Children With Stem Cell Defects, Marrow Failure Syndromes, or Myeloid Leukemia in 1Remission
Brief Title: Busulfan, Antithymocyte Globulin, and Fludarabine Followed By a Donor Stem Cell Transplant in Treating Young Patients With Blood Disorders, Bone Marrow Disorders, Chronic Myelogenous Leukemia in First Chronic Phase, or Acute Myeloid Leukemia in First Remission
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Morton Cowan, Professor, University of California, San Francisco
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000462443; UCSF-01152; UCSF-H411-17802-06
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Congenital Amegakaryocytic Thrombocytopenia; Diamond-blackfan Anemia; Fanconi Anemia; Leukemia; Severe Congenital Neutropenia; Thrombocytopenia
Keywords: thrombocytopenia; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; Diamond-Blackfan anemia; congenital amegakaryocytic thrombocytopenia; Fanconi anemia; severe congenital neutropenia; chronic phase chronic myelogenous leukemia
MeSH Terms: conditions — Congenital amegakaryocytic thrombocytopenia; Anemia, Diamond-Blackfan; Fanconi Anemia; Leukemia; Neutropenia, Severe Congenital, Autosomal Recessive 3; Thrombocytopenia; Leukemia, Myeloid, Chronic-Phase | interventions — Antilymphocyte Serum; Busulfan; fludarabine phosphate; Peripheral Blood Stem Cell Transplantation; Cord Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: anti-thymocyte globulin
Drug: busulfan
Drug: fludarabine phosphate
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Procedure: umbilical cord blood transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as busulfan and fludarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. A donor peripheral blood, bone marrow , or umbilical cord blood transplant may be able to replace blood-forming cells that were destroyed by chemotherapy. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving antithymocyte globulin before the transplant may stop this from happening.

PURPOSE: This phase I/II trial is studying the side effects of busulfan, antithymocyte globulin, and fludarabine when given together with a donor stem cell transplant in treating young patients with blood disorders, bone marrow disorders, chronic myelogenous leukemia in first chronic phase, or acute myeloid leukemia in first remission.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy, in terms of graft rejection at 4 weeks, of a conditioning regimen comprising busulfan, anti-thymocyte globulin, and fludarabine followed by donor stem cell transplantation (SCT) in children with stem cell defects, marrow failure syndromes, chronic myelogenous leukemia in first chronic phase, or acute myeloid leukemia in first remission.
* Determine the pharmacokinetics of busulfan in children undergoing donor SCT.

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine engraftment at 3, 6, 9, and 12 months and mixed chimerism in patients treated with this regimen.
* Determine overall and disease-free survival of patients treated with this regimen.

OUTLINE: Patients receive one of the following cytoreductive regimens:

* Regimen 1 (patients with an HLA genotypic matched sibling donor): Patients receive busulfan IV over 2 hours every 6 hours on days -9 to -6, fludarabine IV on days -5 to -2, and anti-thymocyte globulin (ATG) IV over 10 hours on days -3 to -1.
* Regimen 2 (patients with an HLA closely matched related [not genotypic] or unrelated donor): Patients receive busulfan and fludarabine as in regimen 1, and ATG IV over 10 hours on days -4 to -1.
* Regimen 3 (patients with Fanconi's anemia or severe aplastic anemia with genotypic matched sibling donor): Patients receive fludarabine as in regimen 1 and ATG as in regimen 2.
* Regimen 4 (patients with Fanconi's anemia who have a closely matched related [not genotypic] or unrelated donor): Patients undergo thoracoabdominal irradiation on day -6 and receive fludarabine as in regimen 1 and ATG as in regimen 2.

All patients undergo allogeneic bone marrow, umbilical cord blood, or peripheral blood stem cell transplantation on day 0.

After the completion of study treatment, patients are followed periodically for 20 years.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following hematopoietic disorders:

  * Severe aplastic anemia with marrow aplasia (i.e., absolute neutrophil count < 500/mm^3, platelet and/or red blood cell transfusion dependent), meeting 1 of the following criteria:

    * Closely matched related donor
    * Unresponsive to immunosuppressive therapy within 3 months after follow-up AND alternative matched unrelated donor available
  * Congenital marrow failure syndrome, including any of the following:

    * Primary red blood cell aplasia (Diamond-Blackfan syndrome)
    * Congenital neutropenia (Kostmann's syndrome)
    * Amegakaryocytic thrombocytopenia
  * Hemoglobinopathy including any of the following:

    * β-thalassemia major
    * Sickle cell anemia
  * Severe immunodeficiency disease including any of the following:

    * Chediak-Higashi disease
    * Wiskott-Aldrich syndrome
    * Combined immunodeficiency disease (Nezelof's)
    * Hyperimmunoglobulin M syndrome
    * Bare lymphocyte syndrome
  * Other stem cell defects (e.g., osteopetrosis)
  * Chronic myelogenous leukemia in first chronic phase

    * Not eligible for other ongoing phase II/III studies
  * Acute myeloid leukemia in first remission

    * Not eligible for other ongoing phase II/III studies
  * Inborn errors of metabolism
* No severe combined immunodeficiency disorder
* Available donor, meeting 1 of the following criteria:

  * Related donor matched by high resolution DNA typing at both HLA Drβ1 alleles and ≤ 1 mismatch at the 4 HLA-A and -B alleles
  * Unrelated donor, meeting one of the following criteria:

    * Bone marrow matched by high resolution DNA typing at both HLA Drβ1 alleles and ≤ 1 mismatch by high resolution DNA typing at the 4 HLA-A and -B alleles
    * Umbilical cord blood matched at 4/6 HLA-A, -B, and Drβ1 alleles by high resolution typing with ≥ 1 Drβ1 match and ≥ 3 X 10^7 cells/kg body weight of recipient

PATIENT CHARACTERISTICS:

* See Disease Characteristics
* No active bacterial, viral, or fungal infection
* Cardiac shortening fraction ≥ 27%
* Creatinine clearance ≥ 60 mL/min
* DLCO ≥ 60% of predicted (corrected for anemia/lung volume)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2000-08; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Graft rejection measured by ANC < 500 with no evidence of donor cells in blood or marrow from transplantation to week 4 post transplantation

SECONDARY OUTCOMES:
Toxicity grades 3 or 4 assessed from conditioning through 1 year post transplantation
Engraftment at 1, 3, 6, 9, and 12 months post transplantation
Mixed chimerism at 1, 3, 6, 9, and 12 months post transplantation
Survival measured from the day of first dose of conditioning
Disease-free survival measured from the day of first dose of conditioning

CONTACTS AND LOCATIONS:
Overall Officials: Morton J. Cowan, MD, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Comprehensive Cancer Center, San Francisco, California, United States